CLINICAL TRIAL: NCT00029614
Title: Psychopharmacology of Adolescents With AUD and ADHD
Brief Title: Atomoxetine to Treat Adolescents With Coexisting Alcohol and Other Substance Use Disorder and ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAABUK00301; K24AA000301 (NIH); NIH Grant 5K24AA000301-05
Record Dates: First submitted 2002-01-16; First posted 2002-01-17 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Substance Use Disorders; Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Substance Use
MeSH Terms: conditions — Substance-Related Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of atomoxetine in the treatment of adolescents with coexisting alcohol or substance use disorders and Attention Deficit Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents, ages 13-18
* Meets criteria for alcohol and/or substance use disorder and attention deficit hyperactivity disorder.

Exclusion Criteria:

* Adolescents who are pregnant.
* Have a history of seizure disorder, other neurological or medical disorder for which medication treatment may present a considerable risk.
* History of pervasive development disorder, schizophrenia or other psychotic disorders, organic mental disorders or eating disorders.
* Currently on other psychotropic medications from which discontinuation would present a significant risk.
* A current episode of major depressive disorder or a diagnosis of bipolar disorder.
* Diagnosis of dependence for any substance other than marijuana.
* Adolescents with a full-scale IQ below 80.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-05; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
decrease in ADHD symptoms
decrease in the quantity and frequency of alcohol and other substance use

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G. Bukstein, MD, Principal Investigator — Western Psychiatric Institute and Clinic
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States